CLINICAL TRIAL: NCT02041325
Title: Investigation of the Enhancement of the Response to Hepatitis B Vaccine by Lenalidomide (RevlimidTM, CC-5013) in Plasma Cell Dyscrasias
Brief Title: Investigation of the Enhancement of Response to Hepatitis B Vaccine by Lenalidomide in Plasma Cell Dyscrasias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nikhil Munshi, M.D., Associate Professor of Medicine Harvard Medical School; Physician, Boston VA Research Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: IRB 1831
Record Dates: First submitted 2014-01-14; First posted 2014-01-22 (Estimated); Results first posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: Plasma Cell Disorder
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Lenalidomide; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide (Experimental): Subjects will receive oral CC-5013 (lenalidomide) at 25 mg qd for 7 days prior to and 7 days after the vaccine.
  Interventions: Drug: Lenalidomide
- Placebo (Placebo Comparator): Subjects will receive placebo for 7 days prior to and 7 days after the vaccine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lenalidomide — Subjects will receive oral CC-5013 (lenalidomide) at 25 mg qd for 7 days prior to and 7 days after the vaccine.
  Other Names: CC-5013; Revlimid
  Arms: Lenalidomide
Drug: Placebo — Subjects will receive placebo for 7 days prior to and 7 days after the vaccine.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This is a research study to determine if the study drug lenalidomide will increase the body's immune response, which is the body's response against infections or tumors, to hepatitis B vaccine in patients with plasma cell diseases which include multiple myeloma, monoclonal gammopathy of unknown significance (MGUS) and Waldenström's Macroglobulinemia. It is not a study to see if lenalidomide is an effective treatment for plasma cell disease.

Participants in this study have multiple myeloma or other plasma cell disease and have never been vaccinated with hepatitis B vaccine. One of the effects of the drug lenalidomide is to alter the immune system and thereby increase immune response. It also has some effect against cancer cells; therefore, in theory, it may reduce or prevent the growth of cancer cells.

In this study, one-half of the subjects will be chosen at random to receive the study drug and the other half will take a placebo pill (a sugar pill that looks the same as the real medication). This is a double blind study where neither the subjects nor the investigators know whether the patient receives the study drugs or placebo pills. The effects of the active drug lenalidomide will be compared to the effects of the placebo. The results from this study will be also be compared with a similar but separate study to be done on individuals without known disease.

This study expects to enroll 64 subjects and will be carried out at the Boston VA Healthcare System and the Dana Farber Cancer Institute.

DETAILED DESCRIPTION:
The primary object of this study is to evaluate the effect of CC-5013 on the response to hepatitis B vaccine in myeloma. Secondary objectives include the evaluation of immunologic and functional genomic changes following CC-55013.

This study will be a two-center, randomized, double-blinded, placebo-controlled trial. A single dose of Hepatitis B vaccine will be administered to subjects. CC-5013 or placebo will be administered for 7 days prior to and 7 days after the vaccine. Collection of samples for immune analysis will be performed prior to the initiation of CC-5013 administration, at the time of vaccination, and 7, 14, and 28 days after vaccination. Safety assessment will be performed at each visit.

Primary Endpoint

* Titer of antibodies to hepatitis B virus Secondary Endpoints
* Immune analysis
* Hepatitis B related T cell response
* Safety profile

All the patients should not have a prior response against hepatitis B surface antigen. The study will be comprised of 64 multiple myeloma patients who have not taken any therapeutic agents in the 30 days prior to enrollment in the study. Subjects will be randomly assigned to receive or not receive CC-5013, and all will be vaccinated. The study is designed to detect a biological difference of 50% with an alpha of 0.05 and a beta of 0.8.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age > = 18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Must have confirmed diagnosis of plasma cell disorder.
* Patients with prior thalidomide or CC-5013 (lenalidomide) use are eligible but these agents must have been discontinued at least 4 weeks prior to treatment in this study.
* All previous cancer therapy, including chemotherapy, and dexamethsone must have been discontinued at least 4 weeks prior to treatment in this study. Patients with recent radiation, hormonal therapy and surgery are eligible.
* Patients must not have received prior Hepatitis B vaccination.
* Patient should be negative for antibody against HbSAg.
* ANC >= 1000, Platelets >= 75,000.
* Women of childbearing potential (WCBP) must have a negative urine pregnancy test at screening (Visit 1). In addition, sexually active WCBP must agree to use two of the following adequate forms of contraception throughout the entire study (tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner). A WCBP must agree to have pregnancy tests 4 weeks after her last dose of lenalidomide. Due to the short duration of drug therapy, abstinence would also be a reasonable option.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Concurrent use of other anti-cancer agents or treatments.
* Known HIV, HBV and HCV positivity.
* Clinically significant autoimmune disease.
* Serious intercurrent illness such as active infection requiring IV antibiotics, significant cardiac or pulmonary disease.
* Psychiatric disorder, alcohol or illicit drug use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-04; Primary Completion 2011-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil C Munshi, M.D., Principal Investigator — VA Boston Healthcare System; Harvard Medical School; Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - VA Boston Healthcare System, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide | Placebo
Started | 22 | 16
Completed | 19 | 13
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide | Placebo | Total
Number analyzed (Participants) | 22 | 16 | 38
Age, Continuous [Mean (Full Range); unit: years] | 77 [46 to 90] | 67.5 [47 to 78] | 72.3 [46 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 17 | 10 | 27
Region of Enrollment [Number; unit: Participants]
  United States | 22 | 16 | 38

OUTCOME MEASURES:

1. Primary Outcome: Positive for Hepatitis B Surface Antigen
Description: The number of participants who test positive for the antibody titer against hepatitis B surface antigen (HbSAg).
Time Frame: 6 weeks
Measure: Number; unit: participants
Groups:
- Lenalidomide: Subjects will receive oral CC-5013 (lenalidomide) at 25 mg qd or placebo for 2 weeks.
  Lenalidomide: Subjects will receive oral CC-5013 (lenalidomide) at 25 mg qd or placebo for 2 weeks.
- Placebo: Placebo will be administered for 7 days prior to and 7 days after the vaccine.
  Placebo: Placebo will be administered for 7 days prior to and 7 days after the vaccine.
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 22 | 16
participants | 4 | 3

2. Secondary Outcome: Safety
Description: Number of participants with adverse events as a measure of safety and tolerability
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 22 | 16
participants | 2 | 2

3. Secondary Outcome: Quantity of Subjects With a T-cell Response
Description: Participants who displayed a T cell responses against HbSAg following vaccination
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 22 | 16
participants | 0 | 0

4. Secondary Outcome: Phenotypic Changes
Description: Phenotypic changes in peripheral blood cells following CC-5013 (lenalidomide) administration especially in regards to CD3, CD4, CD8 T cells, and NK and NKT cells.
Time Frame: 6 weeks
Measure: Median (Full Range); unit: cells/cmm
Arm/Group | Lenalidomide | Placebo
Number analyzed (Participants) | 22 | 16
cells/cmm
  Total T cells CD3+ | 851.5 [630 to 1570] | 715 [531 to 1834]
  Helper T cells CD3+/CD4+ | 591 [388 to 1094] | 525 [316 to 1055]
  Cytotoxic T cells CD3+/CD8+ | 296 [77 to 528] | 183 [117 to 1243]
  Natural Killer cells CD56+/CD16+ | 249.5 [98 to 662] | 228 [180 to 418]

ADVERSE EVENTS:
Arm/Group | Lenalidomide | Placebo
Serious Adverse Events (participants affected / at risk) | 2/22 | 2/16
Other Adverse Events (participants affected / at risk) | 0/22 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=22) | Placebo (N=16)
Myocardial Infartion (Cardiac disorders) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ischemic Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No